CLINICAL TRIAL: NCT02304705
Title: Sildenafil in Heart Failure With Reactive Pulmonary Hypertension
Acronym: Sildenafil-HF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty meeting enrollment goal
Sponsor: Maya Guglin (Other)
Responsible Party: Sponsor-Investigator, Maya Guglin, Professor, Clinical Faculty, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-0628-F3R
Record Dates: First submitted 2014-11-26; First posted 2014-12-02 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure With Reactive Pulmonary Hypertension
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo three times per day, orally
  Interventions: Drug: Placebo
- Sildenafil (Active Comparator): Sildenafil 20 mg three times per day, orally
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 20 mg three times daily by mouth for 90 days
  Other Names: Viagra
  Arms: Sildenafil
Drug: Placebo — One capsule three times daily by mouth for 90 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Sildenafil 20mg taken three times a day is effective in the treatment of Heart Failure with Reactive Pulmonary Hypertension. This is a double-blind, placebo controlled trial.

DETAILED DESCRIPTION:
Patients will be screened at the time of a diagnositic Right Heart Catheterization. Patients will be selected based on pressures measured during this procedure, current medications, and current symptoms. At baseline a 6 minute walk test and quality of life questionnaire will be administered. Medical records will be reviewed and results of recent testing will be recorded. Qualifying participants will be randomized to receive 90 days of either placebo or sildenafil 20 mg three times a day. Randomized patients will be followed for safety and efficacy by phone and as otherwise clinically indicated.

At the end of the 90 day treatment period, patients will be evaluated via 6 minute walk, quality of life questionnaire, and other diagnostic tests as clinically indicated. Primary outcome will be change in the 6 minute walk distance. Secondary outcomes will be based on clinically available results such as change in heart pressures measured by right heart catheterization and echocardiogram.

At the end of the treatment period, providers and patients will be unblinded in order to optimize further treatment.

To achieve statistical significance, 64 patients will be enrolled and randomized.

ELIGIBILITY:
Inclusion Criteria:

* Known chronic heart failure appropriately treated with Angiotensin converting enzyme (ACE) inhibitors and beta blockers, unless contraindicated or poorly tolerated
* indication for right heart catheterization
* pulmonary artery mean pressure >25 mmHg
* pulmonary capillary wedge pressure > 15 mmHg
* pulmonary vascular resistance > 3 Wood units

Exclusion Criteria:

* hypersensitivity, allergy, or intolerable side effect to sildenafil
* history of primary pulmonary hypertension, connective tissue disorder, severe chronic obstructive pulmonary disorder (COPD), pulmonary embolism, or left to right shunt
* co-morbidities, limited exercise intolerance:

  * morbid obesity (BMI >40)
  * COPD with oxygen dependence
  * severe peripheral vascular disease with intermittent claudication
  * status post amputation of lower extremity at any level
  * severe degenerative joint disease preventing normal walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maya E Guglin, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guglin M, Rajagopalan N, Anaya P, Charnigo R. Sildenafil in heart failure with reactive pulmonary hypertension (Sildenafil HF) clinical trial (rationale and design). Pulm Circ. 2016 Jun;6(2):161-7. doi: 10.1086/685548. PMID 27252841

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: Sildenafil 20 mg three times per day, orally for 90 days
Period: Overall Study
Arm/Group | Placebo | Sildenafil
Started | 16 | 17
Completed | 12 | 10
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 2 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants had baseline data collected. Only 10 Sildenafil and 12 Placebo had outcome data collects. Several were lost to follow up failures or withdrew either on their own or through PI recommendation.
Groups:
- Placebo: Placebo three times per day, orally
  Placebo: One capsule TID PO for 90 days
- Sildenafil: Sildenafil 20 mg three times per day, orally
  Sildenafil: 20 mg TID PO for 90 days
- Total: Total of all reporting groups
Arm/Group | Placebo | Sildenafil | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 7 | 13 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Tolerance
Description: In a controlled laboratory environment, participants will be asked to walk on a treadmill as fast as they can for 6 minutes. The test will be conducted at baseline and after 90 days of treatment. Data will be presented as the change in distance (in feet) walked in 6 minutes between baseline and treatment.
Time Frame: Baseline and 90 days
Population: Several participants were not analyzed for several reasons including death, failure to follow-up, PI withdrawal or subject withdrawal. In the Sildenafil group, 17 participants were consented while 10 were analyzed. In the Placebo group, 16 subjects were consented and 12 were analyzed.
Measure: Mean (Standard Error); unit: feet
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 12 | 10
feet | 228 (174) | 135 (22)
Statistical Analysis 1: Comparison: Placebo vs Sildenafil; Test type: Superiority; p = .052, t-test, 2 sided

2. Other Pre Specified Outcome: Change in Right Ventricular Function
Description: Right ventricular function will be measured using tricuspid annular plane systolic excursion via two dimensional apical four-chamber echocardiography. Data will be collected at baseline and after 90 days of treatment
Time Frame: Baseline and 90 day
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in Cardiac Output Relative to Body Surface Area (Cardiac Index)
Description: cardiac output will be calculated by multiplying stroke volume by heart rate. Cardiac index will be calculated by dividing cardiac output (Liters/minute) by body surface area (meters squared). Data will be collected at baseline and the end of treatment (90 days)
Time Frame: Baseline and 90 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Pulmonary Vascular Resistance
Description: Pulmonary vascular resistance will be determined by right heart catheterization. Data will be collected at baseline and at the end of treatment (90 days)
Time Frame: Baseline and 90 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Blood Pressure
Description: through standard cuff method, participants will have blood pressure measured to determine systolic and diastolic blood pressure as well as mean arterial pressure. data will be collected at baseline and 90 days.
Time Frame: Baseline and 90 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 90 days from the date of consent until the drug protocol was complete.
Description: Does not differ
Arm/Group | Placebo | Sildenafil
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

LIMITATIONS AND CAVEATS:
There is a real risk that individuals presenting to the cardiology clinics will choose not to participate based on the physical exertion requirement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT02304705/Prot_SAP_000.pdf